CLINICAL TRIAL: NCT04861519
Title: Pivotal, Single-arm Clinical Trial (Prospective Analysis of Retrospective Data) to Assess the Efficacy and Safety of the MedHub AutocathFFR Software Device in Measuring FFR From Digital Angiography Images as a Supportive Aid in the Evaluation and Assessment of Hemodynamically Significant Coronary Artery Disease
Brief Title: Pivotal, Single-arm Clinical Trial to Assess the Efficacy and Safety of the MedHub AutocathFFR Software Device
Acronym: AutocathFFR
Status: Completed | Type: Observational
Sponsor: Medhub Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN-FFR-002
Record Dates: First submitted 2021-04-21; First posted 2021-04-27 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Stable Angina; Unstable Angina; NSTEMI
Keywords: coronary angiography
MeSH Terms: conditions — Angina, Stable; Angina, Unstable; Non-ST Elevated Myocardial Infarction | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- adult subjects who underwent a clinically indicated invasive coronary angiography: adult subjects with stable angina, unstable angina or NSTEM1 who underwent a clinically indicated invasive coronary angiography and on whom invasive FFR has been measured in vessels with coronary lesions.
  Interventions: Other: Collecting invasive FFR measurements.

INTERVENTIONS:
Other: Collecting invasive FFR measurements. — Invasive FFR measurements from the patient's hospital records will be collected.
  Other Names: data collection

SUMMARY:
Prospective (analysis of retrospective data), multi-center, observational, single-arm study. This structure was selected as the "worst case" due to the fact that it represents real life usage of invasive FFR measurement is performed mostly in "gray zone" cases, which are that their severity cannot be determined intuitively and based on the physician eyeball. By using real-world historical data of invasive FFR, the analysis of the obtained data can ensure that the study results are expected to include invasive FFR results that are in the grey zone, when invasive FFR is used in real life and represent the real expected use of the product. Furthermore, the analysis of the data obtained in the studies with these similar devices measuring FFR obtained from angiograms was actually performed in a retrospective manner. That is, although the angiographic images and pressure wire recordings were obtained in real-time, due to the need to mark the vessel in real-time and obtain specific projections during the procedure without which the FFR cannot be calculated, the primary endpoint (sensitivity and specificity) and accuracy were determined in all studies by a post-hoc review by a similar independent QCA core laboratory. The invasive FFR data, as well as the software generated FFR data were reviewed post-hoc by a core laboratory or even at the company.

DETAILED DESCRIPTION:
The proposed study is designed to compare MedHub AutocathFFR measurements obtained from angiograms for the non-invasive determination of the presence of hemodynamically significant coronary lesions. The software device will run on angiograms generated during cardiac catheterization and results will be compared to invasive FFR measurements.

The study is a prospective (analysis of retrospective data), multi-center, observational, single-arm, study.

A total of 308 cases will be enrolled in the study. The study population who represent the target population for this procedure consists of subjects with stable angina, unstable angina or NSTEM1 who underwent a clinically indicated invasive coronary angiography and for whom invasive FFR have been measured in vessels with coronary lesions. For each lesion of interest, a minimum of two 2D angiographic projections, will be obtained. Patients of both genders, all ethnicities, >18 years of age will be recruited to the study. Study cases will be sourced from numerous hospitals in the United States and Israel.

Investigators will screen cases based on the inclusion/exclusion criteria described below. General patient demographics, medical history, concomitant medications, C-arm angiography system used, FFR pressure wire used, etc., will be obtained for each study case.

Subjects with known or suspected coronary artery disease who were scheduled for clinically indicated invasive coronary angiography (ICA) and on whom invasive FFR has been measured in vessels with coronary lesions will comprise the patient population. Coronary angiography will have been performed in a routine fashion in patients with suspected coronary artery disease. When clinically indicated, invasive FFR will have been measured in vessels with coronary lesions of varying severity using a coronary pressure wire and hyperemic stimulus.

The patient's angiographic images will be sent to an independent Quantitative Coronary Arteriography (QCA) Core Laboratory, where they will be processed using the MedHub AutocathFFR device, by independent potential users of the device (i.e., interventional cardiologists). The users will use the diagnostic angiograms and upload them to the AutocathFFR device, to generate the AutocathFFR value. The independent users will be blinded to the software device-generated FFR results and to the invasive FFR measurements. Blinding will be employed in the study because the primary endpoint, i.e., the scored FFR measurements per vessel are subject to bias by device users. Observations in patients with more than 1 study vessel will be presumed independent. The AutocathFFR will not be used for diagnostic or clinical decisions. A detailed standard operating procedure (SOP) for AutoCathFFR computation will be provided to the QCA Core Laboratory.

The AutocathFFR device automatically suggests and marks locations of suspicious narrowing and computes an FFR value for each detected area. The clinician can also select and mark manually locations with suspected narrowing for computing of FFR value. The clinical performance of AutocathFFR device depends only on the uploaded angiograms, on which the AutocathFFR results are presented alongside the viewed blood vessel. There is no need for user interaction with the system during the diagnostic angiography procedure. For example, there is no need to take specific orthogonal projection nor to designate or mark the blood vessels or segments. When the desired coronary artery is viewed on the Cath Lab monitor, the AutocathFFR measurement is automatically shown alongside the viewed vessel, if an area of narrowing is identified in the vessel. Therefore, the use of the AutocathFFR device is seamless with the angiographic imaging procedure and does not require any additional intervention by the cardiologist.

ELIGIBILITY:
Inclusion Criteria:

patient specific:

* Age > 18 years.
* Subjects with stable angina pectoris, unstable angina pectoris or NSTEM1 and in whom invasive FFR was performed to assess a non-culprit stenosis in at least one coronary artery.

Angiographic:

* Subject underwent a clinically indicated Invasive Coronary Angiogram (ICA).
* Subject underwent invasive FFR with IV or intracoronary Adenosine, Adenosine Triphosphate (ATP) or Papaverine used as hyperemic stimulus.

Exclusion Criteria:

Patient Specific:

* Angiogram not obtained on an FDA cleared C-Arm angiography system.
* Invasive FFR not obtained on an FDA cleared FFR catheter tip pressure transducer (a.k.a. pressure wire).
* Vessel size less than 2 mm.
* Subject presents with an acute infarct (STEM1) OR has documented prior STEMI on same side (right/left).
* CTO in target vessel.
* Prior CABG, heart transplant or valve surgery, prior TAVI/TAVR or severe left sided valvular disease.
* Known LVEF ≤45%.
* Arteries supplying akinetic or severe hypokinetic territories if already known based on prior imaging.
* TIMI Grade 2 or lower at baseline.
* Target lesion involves Left Main (stenosis >50%).
* PCI with stent in target vessel in past 12 months, or target vessel involves in-stent restenosis.
* Severe, diffuse disease defined as the presence of diffuse, serial gross luminal irregularities present in the majority of the coronary tree.
* Target coronary vessel provides collaterals to a chronically occluded vessel.

Angiographic:

* Coronary angiography was performed per standard of care at a cine frame rate of at least 7 frames per second.
* Presence of aortic damping.
* Distortion of the waveform.
* A minimum of two different angiographic views for each lesion of interest in the Left Circumflex Artery (LCX), Left Descending Artery (LAD) and in the Right Circumflex Artery (RCA).
* Lesion is not clearly visible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: C-Arm images from adult subjects with stable angina, unstable angina or NSTEM1 who underwent a clinically indicated invasive coronary angiography and on whom invasive FFR has been measured in vessels with coronary lesions.
Sampling Method: Probability Sample
Enrollment: 308 (Actual)
Dates: Start 2021-05-09 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluate the sensitivity and specificity of AutoCathFFR | Up to 2 months
  Co-primary endpoints are the sensitivity and specificity of the dichotomously scored AutocathFFR per vessel compared to the gold standard, invasive FFR measurements, where an FFR ≤ 0.80 is scored "positive" and an FFR > 0.80 is considered "negative".

SECONDARY OUTCOMES:
To assess the accuracy | Up to 2 months
  To assess the accuracy, positive predictive value and negative predictive value and per lesion of the AutocathFFR in correctly diagnosing both positive, as well as negative hemodynamically significant coronary stenosis, using the invasive FFR as the reference standard.
To assess the corelation bwtween invasive FFR and AutoCathFFR | Up to 2 months
  To assess continuously scored AutocathFFR overall correlation with the invasive FFR measurements
To assess the sensitivity and specificity | Up to 2 months
  To assess the sensitivity and specificity of the dichotomously scored AutocathFFR index per lesion.
To assess device success rate | Up to 2 months
  To assess device success, measured as the ratio of completed versus initiated AutocathFFR index calculations.
To assess the Usability of the AutocathFFR | Up to 2 months
  To assess the Usability of the AutocathFFR device, as evaluated using a questionnaire focusing on ease of use and intuitiveness of the system, to be completed by the user (i.e., interventional cardiologists).
Comprehensiveness of the User Manual | Up to 2 months
  Comprehensiveness of the User Manual, to be rated using a questionnaire completed by the user (i.e., interventional cardiologists in the QCA Core Lab)
Device-related adverse events/malfunction | Up to 2 months
  Device-related adverse events/malfunction

CONTACTS AND LOCATIONS:
Locations (3):
- Israel (3):
  - Hillel Yaffe Medical Center, Hadera, Central District
  - Rambam Medical Center, Haifa, North
  - Soroka Medical Center, Beersheba, South